CLINICAL TRIAL: NCT00342771
Title: A Case-Control Study of Prostate Cancer in the Greater Baltimore Area: An Epidemiological Study of Genetic Risk Factors for Prostate Cancer in African-American and Caucasian Males
Brief Title: An Epidemiological Study of Genetic Risk Factors for Prostate Cancer in African-American and Caucasian Males
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905021; 05-C-N021; NCT00556725 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer
Keywords: Tobacco Use; Tumor Biology; Biomarker; Risk Factor; Health Disparity
MeSH Terms: conditions — Prostatic Neoplasms; Tobacco Use

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NCI Maryland pop-based controls: population-based controls
- NCI-Maryland Prostate Cancer Cases: prostate cancer cases

SUMMARY:
This study will examine the association of genetic variants and gene expression patterns with the risk of prostate cancer. There will be (It will include?) genotype analysis of blood DNA from 600 patients with the disease and from 600 healthy people, and there will be a gene expression analysis of prostate tumors. Prostate cancer is a leading cause of death among men in Western countries. It is estimated that 220,000 or more new cases of the disease will occur in the United States during 2004. The disease incidence is rising. About 25% to 30% of the cancers become aggressive. The nonhereditary disease rarely occurs in men who are younger than age 40. There are large differences in incidence by geography and race. The highest rates are seen among African-American men in the United States. Also, although Caucasians have a lower rate of disease incidence and mortality in the United States, the rates among them are high compared with rates in some European countries. The reasons for such differences are not well understood, but both environmental and genetic risk factors are thought to be involved.

Patients ages 40 to 80 years who have had prostate cancer confirmed within the past 6 months, who reside in Baltimore City or adjacent metropolitan counties, and who were born in the United States may be eligible for this study. They will be recruited in collaboration with the Departments of Pathology and Urology at the University of Maryland and the Baltimore Veterans Affairs Medical Center. Those men serving as controls in this study will be identified through the Department of Motor Vehicles database and will be matched by age and race with the patients who have cancer. The study will include 600 participants with prostate cancer and 600 participants in the control group.

Trained interviewers will administer two questionnaires. The primary questionnaire will be used to assess information such as medical and cancer history, tobacco use, current medications, occupational history, family medical history, and socioeconomic status. A supplemental questionnaire will pertain to patients' exposure to risk factors for prostate cancer. It will assess the human body, diet, medical history, family medical history, and sexual history. The section on sexual history will be self-administered.

Patients will undergo collection of blood and urine for various tests. For cancer patients with prostate surgery, there will also be a collection of tissue, to be performed at the time that the prostate gland is scheduled for surgical removal. The pattern of gene expression will be analyzed in low- and high-stage tumors.

There will be no direct benefit from participating in the study, but participants will receive an incentive of up to $75 to participate in the study. No form of treatment is involved in this study. However, it is hoped that the study findings will improve researchers' understanding of prostate cancer biology with respect to the causes of the health variances between African-Americans and Caucasians.

...

DETAILED DESCRIPTION:
We are conducting an epidemiological prostate cancer case-control study in Baltimore, Maryland. Participants will be African American and Caucasian males who reside in Baltimore city and surrounding areas. The study is ongoing and will recruit 1000 prostate cancer cases and 1000 population-based controls. The cases are recruited at two Baltimore hospitals, the Veterans Affairs Medical Center and the University of Maryland Center. Cases will have pathologically confirmed prostate cancer. The population-based controls are identified through the Maryland Department of Motor Vehicle Database, and are frequency-matched by age and race to cases. Enrollment of controls started concurrently with case accrual. The first 12 months of the study constituted a pilot study, during which we evaluated the recruitment procedures. The study involves the administration of two questionnaires and collection of blood from all study subjects. The two questionnaires consist of a main questionnaire and a supplemental questionnaire. The questionnaires evaluate family cancer history, tobacco use, medication, occupational history, socioeconomic status and risk factors for prostate cancer. Fresh-frozen tumor specimens will be obtained from cancer patients if available. The study is supported by an epidemiological infrastructure that has been developed by our resource contractor at the University of Maryland for a lung cancer case-control study. This lung cancer study is ongoing, and the controls that are recruited for the prostate cancer study are joint controls with the lung cancer study. Hence, population-based male controls recruited by our contractor have double eligibility for the concurrent lung and prostate cancer studies. To achieve an age and race matching of cases and controls in the prostate study, we will over-sample male controls in the lung study.

We will test the primary hypothesis that genes and environmental exposures, including infections and medical history, and interactions between those exposures and genetic factors modify prostate cancer susceptibility. As the secondary goal, we will study gene expression profiles of prostate tumors to identify changes in tumor biology that are associated with exposure to genetic and environmental risk factors. It is a focus of this research to identify mechanisms in tumor biology that may cause the aggressive nature of prostate cancer in African American men.

ELIGIBILITY:
* ELIGIBILITY CRITERIA

CASE SUBJECT SELECTION

We will recruit incident cases of pathologically confirmed PCa at all stages of the disease that are age 40 to 90 years. Treatment can be surgery or therapy. The following check list will be used to verify eligibility of a case subject.

ELIGIBILITY CHECK LIST - PROSTATE CANCER CASES

CRITERIA (ALL MUST BE CHECKED):

* Has been diagnosed with prostate cancer within the last two years
* Pathological diagnosis of prostate cancer made at the local hospital pathology department
* Resides in Baltimore City or contiguous metropolitan counties, Anne Arundel and Prince George s counties, Eastern Shore, western and northern Maryland, or adjacent counties in Pennsylvania, Delaware, Virginia, or the Washington Metropolitan area
* Has a residential working phone within his home
* Born in the United States
* Of African-American or Caucasian descent, and age 40 to 90 years
* A non-objection statement by the physician from the hospital where the patient was identified, or listed as the treating physician by the tumor registry or surgical pathology report, to contact the patient
* Is not currently residing in an institution, such as a prison, nursing home, or shelter
* Is not a severely ill patient in the intensive care unit
* Speaks English well enough to be interviewed
* Is able to give informed consent
* Is physically and mentally capable of performing the interview
* Has never been interviewed as a control for this study
* Subject provides informed consent and signs form.

Unwilling Unavailable

SELECTION OF POPULATION-BASED CONTROLS

Population-based controls will be identified through the Department of Motor Vehicles (DMV), and matched on age (5-year intervals), gender and race to cases. Recruitment of controls will start concurrently with case accrual, using the age and race frequency distribution of cancer patients in previous years, but recruitment objectives can be re-assessed to ensure a frequency-matched study. We will exclude controls that do not have a listed home phone number. The following check list will be used to verify eligibility of a control subject.

ELIGIBILITY CHECK LIST - POPULATION-BASED CONTROLS

CRITERIA (ALL MUST BE CHECKED):

* Resides in Baltimore City or contiguous metropolitan counties, Anne Arundel and Prince George s counties, Eastern Shore, western and northern Maryland, or adjacent counties in Pennsylvania, Delaware, Virginia, or the Washington Metropolitan area
* Has a residential working phone within his home
* Born in the United States
* Of African-American or Caucasian descent, and age 40 to 90 years
* Does not have a personal history of cancer other than basal and non-melanomic skin cancer
* Have never had radiation therapy or chemotherapy

Is not currently residing in an institution, such as a prison, nursing home, or shelter

* Speaks English well enough to be interviewed
* Is able to give informed consent
* Is physically and mentally capable of performing the interview
* Has never been interviewed as a control for the study
* Subject provides informed consent and signs form.

Unwilling Unavailable

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is a case-control study with a clinical and a community component. Participants are African- American and Caucasian males who resided in Baltimore city and surrounding areas. The cases were recruited at two Baltimore hospitals, the Veterans Affairs Medical Center and the University of Maryland Medical Center. Cases had pathologically confirmed prostate cancer. The population-based controls were identified through the Maryland Department of Motor Vehicle database.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 2033 (Actual)
Dates: Start 2004-11-08 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Identification of risk factors | After completion of recruitment
  association of tobacco use, obesity, inflammation and anti- inflammatory drugs, sexual activity and sexually transmitted diseases, and ancestral markers with prostate cancer and lethal disease
Identification of disease biomarkers | Ongoing
  association of blood and/or urine-based metabolites, and blood-based immune- inflammation markers with either ancestry, lifestyle factors, prostate cancer, and lethal disease.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Ambs, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - University of Maryland Medical Center, Baltimore, Maryland
  - VA Hospital, Baltimore, Baltimore, Maryland

REFERENCES:
- [Background] DeMarzo AM, Nelson WG, Isaacs WB, Epstein JI. Pathological and molecular aspects of prostate cancer. Lancet. 2003 Mar 15;361(9361):955-64. doi: 10.1016/S0140-6736(03)12779-1. PMID 12648986
- [Background] Roberts WW, Platz EA, Walsh PC. Association of cigarette smoking with extraprostatic prostate cancer in young men. J Urol. 2003 Feb;169(2):512-6; discussion 516. doi: 10.1097/01.ju.0000046160.80804.7f. PMID 12544299
- [Background] Hoffman RM, Gilliland FD, Eley JW, Harlan LC, Stephenson RA, Stanford JL, Albertson PC, Hamilton AS, Hunt WC, Potosky AL. Racial and ethnic differences in advanced-stage prostate cancer: the Prostate Cancer Outcomes Study. J Natl Cancer Inst. 2001 Mar 7;93(5):388-95. doi: 10.1093/jnci/93.5.388. PMID 11238701